CLINICAL TRIAL: NCT02205203
Title: Expanding Access to Therapy for Childhood Anxiety Disorders Via Smart Phones - RCT
Brief Title: Youth Mayo Clinic Anxiety Coach Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stephen Whiteside (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Stephen Whiteside, Professor of Psychology, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13-000288 - RCT; R34MH100468 (NIH)
Record Dates: First submitted 2014-07-29; First posted 2014-07-31 (Estimated); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Anxiety
Keywords: Anxiety; Social Anxiety; Social Phobia; Separation Anxiety; Generalized Anxiety; GAD; Phobia; Panic; Agoraphobia; Obsessive Compulsive Disorder; OCD; Child; Adolescent; Smartphone; Teen; Youth
MeSH Terms: conditions — Anxiety Disorders; Phobia, Social; Anxiety, Separation; Generalized Anxiety Disorder; Phobic Disorders; Agoraphobia; Obsessive-Compulsive Disorder | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Face-to-Face w/ Anxiety Coach (FTF-AC) (Active Comparator): In this condition therapists will provide 6 to 12 50-minute, face-to-face therapy sessions using Mayo Clinic Anxiety Coach. The sessions are expected to initially occur weekly and be within the office although the therapist can leave the office to conduct exposure. The therapist is expected to utilize Anxiety Coach within the session, encourage the patient to use the application to complete homework, and review progress in-session via the web-based portal.
  Interventions: Device: Mayo Clinic Anxiety Coach
- Treatment as Usual (TAU) (Experimental): In the TAU condition therapists provide treatment consistent with their orientation and clinical judgment. Previous research suggests that TAU will include supportive therapy, relaxation, and cognitive restructuring. The format of treatment will be 6 to 12, 50-minute, face-to-face therapy sessions in the therapist's office, with flexibility to leave the office (e.g., for exposure). Therapists can communicate with patients between sessions (e.g., phone calls), as long as this medium is not the primary mode of treatment.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Device: Mayo Clinic Anxiety Coach — Mayo Clinic Anxiety Coach is a smartphone application based on cognitive-behavioral treatment for anxiety disorders (i.e., exposure-based therapy) that can be used as 1) a stand-alone treatment requiring minimal provider contact, and 2) an augmentation of face-to-face treatment that increases clinician fidelity and patient adherence to evidence-based treatment. The design of Anxiety Coach is based on evidence and theory suggesting that information and communication technologies (ICTs) are well-suited for encouraging behavior change through 1) scheduled reminders to engage in therapeutic exercises, 2) point of performance support, 3) individually tailored information, 4) real-time symptom assessment, and 5) readily accessible asynchronous communication.
  Arms: Face-to-Face w/ Anxiety Coach (FTF-AC)
Other: Treatment as Usual — In the TAU condition therapists provide treatment consistent with their orientation and clinical judgment. Previous research suggests that TAU will include supportive therapy, relaxation, and cognitive restructuring. The format of treatment will be 6 to 12, 50-minute, face-to-face therapy sessions in the therapist's office, with flexibility to leave the office (e.g., for exposure).
  Arms: Treatment as Usual (TAU)

SUMMARY:
This research study aims to test the feasibility and effectiveness of using the Mayo Clinic Anxiety Coach smartphone app as an addition to traditional therapy for the treatment of anxiety disorders in youth, particularly those youth who may have limited access to mental health treatment in the traditional clinical setting.

DETAILED DESCRIPTION:
60 therapists in underserved areas will treat children with anxiety disorders in one of three conditions (treatment as usual, Anxiety Coach with face-to-face therapy, or Anxiety Coach with minimal direct contact) to determine the feasibility of using of Anxiety Coach to increase the frequency of exposure and improve outcomes with varying degrees of face-to-face contact (N = 60 patients).

ELIGIBILITY:
Inclusion Criteria:

1. Age 7 to 17
2. Primary diagnosis of:

   1. social phobia,
   2. separation anxiety disorder,
   3. panic disorder with and without agoraphobia,
   4. specific phobia, or
   5. obsessive compulsive disorder
3. A parent or other primary care giver available to participate with the child in all assessment and treatment activities
4. Estimated average intelligence
5. English speaking

Exclusion Criteria:

1. History of and/or current diagnosis of:

   1. psychosis,
   2. autism,
   3. bipolar disorder,
   4. mental retardation,
   5. oppositional defiant disorder,
   6. PTSD,
   7. selective mutism, or
   8. major depressive disorder
2. Current suicidality or recent suicidal behavior
3. Parent to be involved in study who is unable to adequately participate due to intellectual or psychiatric difficulties
4. Starting or changing the dosage of a psychiatric medication in the last two months

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 145 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Mean change from Baseline in Pediatric Anxiety Rating Scale (PARS) at Treatment Completion | Within 5 working days of Treatment Completion
  The Pediatric Anxiety Rating Scale (PARS) is an interview-based tool used to assess for the presence and severity of anxiety symptoms in children and adolescents utilizing parental and youth input to guide clinician ratings.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Whiteside, Ph.D., L.P., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Whiteside SPH, Sawchuk NR, Brennan E, Lebow JR, Sawchuk CN, Biggs BK, Dammann JE, Tiede MS, Hofschulte DR, Reneson-Feeder S, Cunningham M, Allison ML. Using session recordings to understand the content of community-based treatment for childhood anxiety disorders and response to technology-based training. J Clin Psychol. 2023 Oct;79(10):2251-2269. doi: 10.1002/jclp.23537. Epub 2023 May 20. PMID 37209422